CLINICAL TRIAL: NCT04757324
Title: The Influence of Breast Milk and Breastfeeding Education Given in the Antenatal Period on Breastfeeding Success and Breastfeeding Self-efficacy: Randomize Control Trials
Brief Title: Breast Milk and Breastfeeding Education Given in the Antenatal Period
Acronym: BSES-SF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Collaborators: Balikesir University (Other)
Responsible Party: Principal Investigator, Rukiye Öztürk, M.Sc., Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Breastfeeding Education
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Breastfeeding
Keywords: Breastfeeding success; Breastfeeding education; Breastfeeding self-efficacy perception; Breast milk; Antenatal period
MeSH Terms: conditions — Breast Feeding | interventions — Prenatal Education

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education arm (Experimental): Breastfeeding training was given to the training arm
  Interventions: Other: breastfeeding education
- control arm (No Intervention): Breastfeeding training not given to control arm

INTERVENTIONS:
Other: breastfeeding education
  Other Names: antenatal education
  Arms: education arm

SUMMARY:
We aimed to examine the influence of breast milk and breastfeeding education given in the ante-natal period on LATCH score and breastfeeding self-efficacy score.

DETAILED DESCRIPTION:
Practices for increasing breastfeeding self-efficacy are of vital importance and they increase the level of breastfeeding self-efficacy. Breast milk and breastfeeding educations have given in the ante-natal period are another way of increasing the success of breastfeeding.

In this experimental investigation, 80 pregnant women who attended a baby-friendly hospital were randomly assigned to the education (n = 40) or control (n = 40) groups. The pregnant women in the intervention group received 4 hours of human milk and breastfeeding educational sessions along with routine care and furthermore, a brochure prepared by the researcher was given. All women whose estimated delivery date had approximated were questioned about whether they had given birth or not, and the sociodemographic data form, the LATCH Breastfeeding Assessment Tool and the Breastfeeding Self-efficacy Scale-short form were applied to the subjects in the education and the control group by visiting them at home when the post-partum first week had been completed.

ELIGIBILITY:
inclusion criteria Being above 18 years of age, Having completed the 26th gestational week (At training phase), Having no problem with vision and hearing, Having no disease that can prevent breastfeeding, Having a pregnancy with no risk, Having no systemic disease, Planning to breastfeed after birth

excusion criteria the mother stops researching. treating the baby in neonatal intensive care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 67 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in self-efficacy on the 70 points Breastfeeding Self-efficacy Scale-short form at week 1 | baseline and week 1
Change from baseline in LATCH score on the 70 points LATCH Breastfeeding Assessment Toolform at week 1 | baseline in week 1
  breastfeeding success

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozturk R, Ergun S, Ozyazicioglu N. Effect of antenatal educational intervention on maternal breastfeeding self-efficacy and breastfeeding success: a quasi-experimental study. Rev Esc Enferm USP. 2022 Apr 4;56:e20210428. doi: 10.1590/1980-220X-REEUSP-2021-0428. eCollection 2022. PMID 35377385